CLINICAL TRIAL: NCT06199336
Title: A Phase I/II, Randomized, Double-blind, Placebo, and Active Controlled Clinical Study to Evaluate the Safety, Tolerability, Immunogenicity, and Preliminary Efficacy of JHM03 in Subjects With Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: JHM BioPharma (Tonghua) Co. , Ltd. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JHM03-CT101
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-04

CONDITIONS: Moderate to Severe Glabellar Lines
Keywords: Recombinant Botulinum Toxin Type A, Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Placebo and active controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment Group (Experimental): Single injection with JHM03 in glabellar lines
  Interventions: Biological: JHM03
- Active-Controlled Group (Active Comparator): Single injection with BOTOX® in glabellar lines
  Interventions: Biological: BOTOX®
- Placebo-Controlled Group (Placebo Comparator): Single injection with Placebo in glabellar lines.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: JHM03 — Single treatment, intramuscularly injected into five sites. The total injection volume is 0.5 ml,0.1 ml per site.
  Arms: Treatment Group
Biological: BOTOX® — Single treatment,intramuscularly injected into five sites.The total injection volume is 0.5 ml,0.1 ml per site.
  Arms: Active-Controlled Group
Biological: Placebo — Single treatment,intramuscularly injected into five sites.The total injection volume is 0.5 ml,0.1 ml per site.
  Arms: Placebo-Controlled Group

SUMMARY:
This is a phase 1/2, multicenter, randomized, double-blind, active-controlled and placebo-controlled study to evaluate safety, immunogenicity and efficacy of JHM03 for the treatment of moderate to severe glabellar lines in male and female subjects of Chinese origin. The purpose of this study was to observe efficacy and safety of JHM03 compared with placebo and BOTOX® in moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 65 years of age.
2. Moderate to severe glabellar lines at maximum frown at baseline.

Exclusion Criteria:

1. Previous use of any botulinum toxin within 6 months prior to screening, or plan to use any botulinum toxin during the study.
2. Use of medications that affect neuromuscular transmission within 4 weeks prior to screening, such as muscle relaxant,aminoglycoside antibiotics,anticholinergic drugs,benzodiazepines,etc.
3. Suffering from any neurological disorders that increase the risk of exposure to botulinum toxin type A, including peripheral motor nerve diseases (such as amyotrophic lateral sclerosis and motor neuropathy), as well as neuromuscular junction diseases (such as Lambert-Eaton syndrome and myasthenia gravis).
4. Known allergy or hypersensitivity to any component of the study products.
5. Use of any non-steroid anti-inflammatory drug or anticoagulant within 1 week prior to study treatment.
6. History of alcohol or drug abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Phase1 | Within 28 days
  The incidence rate of adverse events and severe adverse events within 28 days after injection;
Phase2 | within 4 weeks
  Percentage of Subjects as Responders in the Investigator's live assessment (Using 4-point Photographic Scale) and the subject's self assessment of Glabellar Lines at Maximum Frown.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Second Provincial General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No